CLINICAL TRIAL: NCT04483193
Title: Reliability of Extended Duplex Ultrasound for Diagnosis of Proximal Deep Vein Thrombosis Performed by General Intensive Care Unit Nurses in the Critically Ill Patients
Brief Title: Reliability of Duplex Ultrasound for Diagnosis of Deep Vein Thrombosis Performed by Nurses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Emergency Medical Service of the Central Bohemian Region, Czech Republic (Other)
Collaborators: Masaryk Hospital Usti nad Labem (Other)
Responsible Party: Principal Investigator, Roman Skulec, Principal investigator, Masaryk Hospital Usti nad Labem
Other Study IDs: 284/36
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Ultrasound
MeSH Terms: interventions — Ultrasonography, Doppler, Duplex

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients: Critically ill patients hospitalised at the intensive care unit.
  Interventions: Diagnostic Test: Duplex ultrasound

INTERVENTIONS:
Diagnostic Test: Duplex ultrasound — Point-of-Care compression ultrasound test combined with colour doppler imaging in the range from the groin to the popliteal region of both lower extremities.

SUMMARY:
The purpose of this study is to assess validity of extended duplex ultrasound examination for diagnosis of proximal deep vein thrombosis performed by general intensive care unit nurses in the critically ill patients.

DETAILED DESCRIPTION:
Critically ill patients hospitalized in the intensive care unit are in increased risk of proximal deep vein thrombosis despite thromboprophylactic measures. Diagnostic method of the first choice is Point-of-Care ultrasound examination. This method is usually performed by a trained intensive care physician. However, if this examination could be performed by trained nurses, its availability would be greatly increased. The results of the investigator's pilot study showed that general nurses are able to diagnose proximal deep vein thrombosis in critically ill patients by compression ultrasound test with a sensitivity of 88,9 % and a specificity of 99 %. Before implementation of this examination into the optional competencies of general nurses, the results need to be confirmed in a larger group of patients. This is the goal of proposed clinical study.

In this prospective observational study, the patients will be investigated by extended duplex ultrasound (compression ultrasound test combined with colour doppler imaging in the range from the groin to the popliteal region) by a trained nurse and on the same day, the examination will be repeated by a trained physician - intensivist. The results of the examinations of each patient will be blinded until both tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients
* Critically ill patients hospitalised in the intensive care unit for more than 72 hours

Exclusion Criteria:

* Known deep vein thrombosis
* Contraindication of ultrasound examination
* Refusal of ultrasound examination by patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Validity of duplex ultrasound | Comparison of two examinations performed with a maximum interval of 24 hours.
  Validity of duplex ultrasound examination performed by a trained general intensive care nurses when compared with the examination performed by a trained physician - intensivist, specialist in Point-of-Care ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Skulec, MD, PhD, Principal Investigator — Masaryk Hospital Usti nad Labem
Locations (1):
- Masaryk Hospital Usti nad Labem, Ústí nad Labem, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skulec R, Kohlova A, Miksova L, Cerny V. The reliability of ultrasound compression test performed by general ICU nurses in the critically ill patients: A preliminary prospective clinical study. Eur J Intern Med. 2020 Jun;76:130-131. doi: 10.1016/j.ejim.2020.03.007. Epub 2020 Mar 23. No abstract available. PMID 32216998